CLINICAL TRIAL: NCT00974350
Title: A Double-Blind, Placebo-Controlled, Pharmacodynamic and Pharmacokinetic Dose Response Study of SABER-Bupivacaine Instilled Into the Wound in Patients Undergoing Open Inguinal Hernia Repair
Brief Title: A Safety and Efficacy Study of SABER®-Bupivacaine for Pain Following Hernia Repair
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Durect (Industry)
Collaborators: Nycomed (Industry)
Responsible Party: Dmitri Lissin, MD, Sr. Director Clinical Research, Durect Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLIN803-006-0006
Record Dates: First submitted 2009-09-08; First posted 2009-09-10 (Estimated); Results first posted 2021-05-05 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Postoperative Pain; Hernia; Surgery
Keywords: Post-operative pain; hernia surgery; opioid
MeSH Terms: conditions — Pain, Postoperative; Hernia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: SABER-Bupivacaine (Experimental): 2.5 mL SABER-Bupivacaine/Once
  Interventions: Drug: SABER-Bupivacaine
- Group 2: SABER-Bupivacaine (Experimental): 5.0 mL SABER-Bupivacaine/Once
  Interventions: Drug: SABER-Bupivacaine
- Group 3: SABER-Placebo (Placebo Comparator): 2.5 mL or 5.0 mL SABER-Placebo/Once
  Interventions: Drug: SABER-Placebo

INTERVENTIONS:
Drug: SABER-Bupivacaine — Injectable Extended Release Solution; 2.5 mL SABER-Bupivacaine/Once
  Arms: Group 1: SABER-Bupivacaine
Drug: SABER-Bupivacaine — Injectable Extended Release Solution; 5.0 mL SABER-Bupivacaine/Once
  Other Names: POSIMIR® bupivacaine solution
  Arms: Group 2: SABER-Bupivacaine
Drug: SABER-Placebo — Injectable Solution; 2.5 or 5.0 mL SABER-Placebo/Once
  Arms: Group 3: SABER-Placebo

SUMMARY:
This is a research study testing SABER-Bupivacaine (an experimental pain-relieving medication). SABER-Bupivacaine is designed to continuously deliver bupivacaine, a common local anesthetic, for a few days in order to treat local post-surgical pain. This study is testing SABER-Bupivacaine in people having surgery to repair a hernia.

The purpose of the study is to measure and compare the safety (side effects), tolerability (ability to tolerate), and efficacy (how well it works) of two different volumes of SABER-Bupivacaine with SABER-Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 to 65 years of age, scheduled for hernia repair surgery
* Patients must be in good health prior to study participation
* Patients must have blood pressure within normal range or with Stage 1 high blood pressure
* Male and female patients must agree to use medically acceptable method of contraception throughout the entire trial period and for 1 week after the trial is completed
* Patients must refrain from strenuous activities and avoid changes to prescribed exercise levels throughout the course of the trial
* Ability to read, understand, communicate, and voluntarily sign the informed consent form prior to any trial specific procedures

Exclusion Criteria:

* Patients with previous abdominal surgery scar tissue
* Patients with clinically significant abnormalities of any body system unrelated to the disease under study
* Connective tissue disorders
* Patients who are pregnant or lactating
* Current or regular use of analgesic medication for other indications
* Patients with current or regular use of antidepressants or monoamine oxidase inhibitors at screening
* Use of any drugs or medication that may interfere with the study and its results
* Patients with known hypersensitivity to the study drugs or their components
* Patients with known or suspected alcohol abuse or illicit drug use
* Participation in another clinical trial at the same time or within 30 days of this trial
* Patient is unwilling to comply with the study procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2007-01; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitri Lissin, MD, Study Director — Durect
Locations (5):
- Australia (4):
  - Cairns, Queensland
  - Sunnybank, Queensland
  - Port Lincoln, South Australia
  - Ringwood East, Victoria
- Hamilton, New Zealand

REFERENCES:
- [Result] Hadj A, Hadj A, Hadj A, Rosenfeldt F, Nicholson D, Moodie J, Turner R, Watts R, Fletcher I, Abrouk N, Lissin D. Safety and efficacy of extended-release bupivacaine local anaesthetic in open hernia repair: a randomized controlled trial. ANZ J Surg. 2012 Apr;82(4):251-7. doi: 10.1111/j.1445-2197.2011.05754.x. Epub 2011 Jun 24. PMID 22510183

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: SABER-Bupivacaine: 2.5 mL SABER-Bupivacaine/Once
  SABER-Bupivacaine: Injectable Extended Release Solution; 2.5 mL SABER-Bupivacaine(330 mg)/Once
- Group 2: SABER-Bupivacaine: 5.0 mL SABER-Bupivacaine/Once
  SABER-Bupivacaine: Injectable Extended Release Solution; 5.0 mL SABER-Bupivacaine(660 mg)/Once
- Group 3: SABER-Placebo: 2.5 mL or 5.0 mL SABER-Placebo/Once
  SABER-Placebo: Injectable Solution; 2.5 or 5.0 mL SABER-Placebo/Once (SABER-Placebo 2.5 mL or 5.0 mL, as randomly assigned)
Period: Overall Study
Arm/Group | Group 1: SABER-Bupivacaine | Group 2: SABER-Bupivacaine | Group 3: SABER-Placebo
Started | 45 | 47 | 32
Completed | 42 | 47 | 31
Not Completed | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Population: safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: SABER-Bupivacaine | Group 2: SABER-Bupivacaine | Group 3: SABER-Placebo | Total
Number analyzed (Participants) | 44 | 47 | 32 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (11.82) | 48.6 (13.04) | 50.3 (9.26) | 48.11 (11.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 4
  Male | 42 | 45 | 32 | 119
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.5 (3.74) | 26.3 (2.92) | 26.9 (3.68) | 26.55 (3.41)

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity on Movement
Description: Pain intensity on movement normalized AUC over the time period 1 to 72 hours post-surgery. Data on pain intensity were collected using a 0 to 10 NRS with scores ranging from 0 (no pain) to 10 (worst pain possible). The AUC is computed for each patient using the standard trapezoidal rule and normalised by dividing by the time interval over which it is computed. This normalisation converts the AUC to the natural pain scale (NRS 0-10) to allow for better translation of the clinical treatment effect magnitude.
Time Frame: 1 to 72 hours post-dose
Population: ITT population (patients with data available)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Group 2: SABER-Bupivacaine: 5.0 mL SABER-Bupivacaine /Once
  SABER-Bupivacaine: Injectable Extended Release Solution; 5.0 mL SABER-Bupivacaine(660 mg)/Once
Arm/Group | Group 1: SABER-Bupivacaine | Group 2: SABER-Bupivacaine | Group 3: SABER-Placebo
Number analyzed (Participants) | 43 | 47 | 32
score on a scale | 3.4 (0.26) | 2.7 (0.25) | 3.9 (0.29)
Statistical Analysis 1: Comparison: Group 2: SABER-Bupivacaine vs Group 3: SABER-Placebo; Pain Intensity on Movement AUCs1-72 hours Including Pain Assessed Upon Taking Opioid Rescue - ITT; Test type: Superiority; p = 0.0031, ANOVA; LS Mean difference from SABER-Placebo; LS Mean Difference = -1.14, 95% CI 2-sided [-1.84 to -0.44], Standard Error of Mean 0.353

2. Primary Outcome: Proportion (Percent) of Patients Using Supplemental Opioids
Time Frame: 0 to 14 days post-dose
Population: ITT population (patients with data available)
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: SABER-Bupivacaine | Group 2: SABER-Bupivacaine | Group 3: SABER-Placebo
Number analyzed (Participants) | 43 | 47 | 32
Participants | 31 | 25 | 23
Statistical Analysis 1: Comparison: Group 2: SABER-Bupivacaine vs Group 3: SABER-Placebo; Proportion of Patients Not Taking Any Supplemental Opioid Analgesic Medication; Test type: Superiority; p = 0.0909, Cochran-Mantel-Haenszel; Stratified by pooled study sites

3. Secondary Outcome: Pain Intensity
Description: Pain intensity AUC over the time period of 1 to 48 hours. Data on pain intensity were collected using a 0 to 10 NRS with scores ranging from 0 (no pain) to 10 (worst pain possible). The AUC is computed for each patient using the standard trapezoidal rule and normalised by dividing by the time interval over which it is computed. This normalisation converts the AUC to the natural pain scale (NRS 0-10) to allow for better translation of the clinical treatment effect magnitude.
Time Frame: 1 to 48 hours post-dose
Population: ITT population (patients with data available)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Group 1: SABER-Bupivacaine | Group 2: SABER-Bupivacaine | Group 3: SABER-Placebo
Number analyzed (Participants) | 43 | 47 | 32
score on a scale | 3.4 (0.26) | 2.8 (0.26) | 4.1 (0.30)

4. Secondary Outcome: Treatment Satisfaction
Description: Modified Brief Pain Inventory -An overall assessment of treatment satisfaction was made using 6 point verbal rating scale (very dissatisfied, dissatisfied, slightly dissatisfied, slightly satisfied, satisfied, very satisfied).
Time Frame: 1 to 5 days post-dose
Population: ITT population (patients with data available)
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: SABER-Bupivacaine | Group 2: SABER-Bupivacaine | Group 3: SABER-Placebo
Number analyzed (Participants) | 42 | 47 | 30
Participants
  Day 1: number analyzed (Participants) | 42 | 45 | 29
  Day 1: Very Dissatisfied | 2 | 2 | 0
  Day 1: Dissatisfied | 1 | 0 | 2
  Day 1: Slightly Dissatisfied | 1 | 2 | 0
  Day 1: Slightly Satisfied | 2 | 4 | 4
  Day 1: Satisfied | 15 | 16 | 12
  Day 1: Very Satisfied | 21 | 21 | 11
  Day 2: number analyzed (Participants) | 42 | 43 | 30
  Day 2: Very Dissatisfied | 0 | 0 | 1
  Day 2: Dissatisfied | 1 | 0 | 0
  Day 2: Slightly Dissatisfied | 1 | 2 | 2
  Day 2: Slightly Satisfied | 4 | 3 | 4
  Day 2: Satisfied | 15 | 19 | 12
  Day 2: Very Satisfied | 21 | 19 | 11
  Day 3: number analyzed (Participants) | 42 | 45 | 28
  Day 3: Very Dissatisfied | 0 | 0 | 0
  Day 3: Dissatisfied | 0 | 0 | 0
  Day 3: Slightly Dissatisfied | 0 | 0 | 1
  Day 3: Slightly Satisfied | 3 | 2 | 2
  Day 3: Satisfied | 13 | 23 | 14
  Day 3: Very Satisfied | 26 | 20 | 11
  Day 4: number analyzed (Participants) | 38 | 44 | 29
  Day 4: Very Dissatisfied | 0 | 0 | 0
  Day 4: Dissatisfied | 0 | 0 | 1
  Day 4: Slightly Dissatisfied | 0 | 0 | 0
  Day 4: Slightly Satisfied | 2 | 1 | 3
  Day 4: Satisfied | 18 | 21 | 12
  Day 4: Very Satisfied | 18 | 22 | 13
  Day 5: number analyzed (Participants) | 39 | 42 | 27
  Day 5: Very Dissatisfied | 0 | 0 | 0
  Day 5: Dissatisfied | 0 | 0 | 0
  Day 5: Slightly Dissatisfied | 1 | 0 | 1
  Day 5: Slightly Satisfied | 1 | 1 | 1
  Day 5: Satisfied | 16 | 17 | 11
  Day 5: Very Satisfied | 21 | 24 | 14

5. Secondary Outcome: Supplemental Opioid Use
Time Frame: 0 to 14 days post-dose
Population: ITT population (patients with data available)
Measure: Mean (Standard Deviation); unit: Total morphine equivalent dose (mg)
Arm/Group | Group 1: SABER-Bupivacaine | Group 2: SABER-Bupivacaine | Group 3: SABER-Placebo
Number analyzed (Participants) | 43 | 47 | 32
Total morphine equivalent dose (mg) | 17.7 (25.36) | 12.5 (17.63) | 38.4 (60.24)

6. Secondary Outcome: Mean Function Activities (Modified Brief Pain Inventory)
Description: In past 24 hours, pain interfered with ability to function or perform activity (0-10 numeric scale, 0=no interference)
Time Frame: 1 to 5 days post-dose
Population: ITT population (patients with data available)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1: SABER-Bupivacaine | Group 2: SABER-Bupivacaine | Group 3: SABER-Placebo
Number analyzed (Participants) | 43 | 47 | 32
score on a scale
  get out of bed (Day 1): number analyzed (Participants) | 42 | 44 | 28
  get out of bed (Day 1) | 3.2 (2.56) | 2.7 (2.63) | 4.6 (3.49)
  get out of bed (Day 2): number analyzed (Participants) | 42 | 43 | 30
  get out of bed (Day 2) | 3.0 (2.37) | 2.4 (1.88) | 3.0 (2.50)
  get out of bed (Day 3): number analyzed (Participants) | 42 | 45 | 28
  get out of bed (Day 3) | 2.5 (2.09) | 1.5 (1.71) | 2.1 (2.01)
  get out of bed (Day 4): number analyzed (Participants) | 38 | 44 | 29
  get out of bed (Day 4) | 1.7 (1.88) | 1.1 (1.27) | 1.9 (2.12)
  get out of bed (Day 5): number analyzed (Participants) | 39 | 42 | 26
  get out of bed (Day 5) | 1.7 (1.83) | 1.1 (1.33) | 1.4 (1.60)
  Ability to walk (Day 1): number analyzed (Participants) | 41 | 44 | 27
  Ability to walk (Day 1) | 3.5 (2.76) | 2.7 (2.74) | 3.9 (3.14)
  Ability to walk (Day 2): number analyzed (Participants) | 42 | 43 | 30
  Ability to walk (Day 2) | 2.8 (2.25) | 2.3 (2.09) | 2.3 (2.35)
  Ability to walk (Day 3): number analyzed (Participants) | 42 | 45 | 28
  Ability to walk (Day 3) | 2.5 (2.02) | 1.4 (1.62) | 1.5 (1.77)
  Ability to walk (Day 4): number analyzed (Participants) | 38 | 44 | 29
  Ability to walk (Day 4) | 2.0 (1.90) | 1.0 (1.29) | 1.7 (2.45)
  Ability to walk (Day 5): number analyzed (Participants) | 39 | 42 | 26
  Ability to walk (Day 5) | 1.8 (1.89) | 1.3 (1.47) | 1.3 (1.46)
  Ability To Interact With Visitors (Day 1): number analyzed (Participants) | 42 | 45 | 29
  Ability To Interact With Visitors (Day 1) | 1.1 (2.08) | 0.7 (1.32) | 1.4 (1.59)
  Ability To Interact With Visitors (Day 2): number analyzed (Participants) | 42 | 43 | 30
  Ability To Interact With Visitors (Day 2) | 1.0 (1.56) | 1.0 (1.62) | 1.1 (1.31)
  Ability To Interact With Visitors (Day 3): number analyzed (Participants) | 42 | 45 | 28
  Ability To Interact With Visitors (Day 3) | 0.7 (1.22) | 0.4 (0.84) | 0.6 (0.63)
  Ability To Interact With Visitors (Day 4): number analyzed (Participants) | 38 | 44 | 29
  Ability To Interact With Visitors (Day 4) | 0.7 (1.33) | 0.4 (0.73) | 0.5 (1.21)
  Ability To Interact With Visitors (Day 5): number analyzed (Participants) | 39 | 42 | 27
  Ability To Interact With Visitors (Day 5) | 0.5 (1.17) | 0.4 (0.74) | 0.3 (0.61)
  Ability To Fall Asleep (Day 1): number analyzed (Participants) | 42 | 45 | 29
  Ability To Fall Asleep (Day 1) | 2.7 (2.37) | 2.0 (2.31) | 2.6 (2.09)
  Ability To Fall Asleep (Day 2): number analyzed (Participants) | 42 | 43 | 30
  Ability To Fall Asleep (Day 2) | 2.0 (2.25) | 1.3 (1.61) | 1.8 (1.92)
  Ability To Fall Asleep (Day 3): number analyzed (Participants) | 42 | 45 | 28
  Ability To Fall Asleep (Day 3) | 1.5 (1.61) | 0.9 (1.14) | 1.2 (1.31)
  Ability To Fall Asleep (Day 4): number analyzed (Participants) | 38 | 44 | 29
  Ability To Fall Asleep (Day 4) | 1.4 (2.03) | 0.6 (1.14) | 1.3 (2.21)
  Ability To Fall Asleep (Day 5): number analyzed (Participants) | 39 | 42 | 27
  Ability To Fall Asleep (Day 5) | 1.1 (1.52) | 0.5 (0.74) | 0.8 (1.45)
  Ability To Stay Asleep (Day 1): number analyzed (Participants) | 42 | 45 | 29
  Ability To Stay Asleep (Day 1) | 2.6 (2.49) | 2.2 (2.58) | 2.1 (2.28)
  Ability To Stay Asleep (Day 2): number analyzed (Participants) | 42 | 43 | 30
  Ability To Stay Asleep (Day 2) | 2.0 (2.26) | 1.4 (1.79) | 1.8 (2.01)
  Ability To Stay Asleep (Day 3): number analyzed (Participants) | 42 | 45 | 28
  Ability To Stay Asleep (Day 3) | 1.4 (1.67) | 0.7 (1.01) | 1.2 (1.50)
  Ability To Stay Asleep (Day 4): number analyzed (Participants) | 38 | 44 | 29
  Ability To Stay Asleep (Day 4) | 1.2 (1.71) | 0.5 (0.90) | 1.3 (2.33)
  Ability To Stay Asleep (Day 5): number analyzed (Participants) | 39 | 42 | 27
  Ability To Stay Asleep (Day 5) | 1.1 (1.50) | 0.7 (0.92) | 0.7 (1.43)
  Ability To Eat (Day 1): number analyzed (Participants) | 42 | 45 | 29
  Ability To Eat (Day 1) | 1.2 (1.89) | 0.4 (0.94) | 0.9 (1.58)
  Ability To Eat (Day 2): number analyzed (Participants) | 42 | 43 | 30
  Ability To Eat (Day 2) | 0.9 (1.61) | 0.3 (0.72) | 0.5 (1.04)
  Ability To Eat (Day 3): number analyzed (Participants) | 42 | 45 | 28
  Ability To Eat (Day 3) | 0.5 (1.06) | 0.2 (0.55) | 0.4 (1.19)
  Ability To Eat (Day 4): number analyzed (Participants) | 38 | 44 | 29
  Ability To Eat (Day 4) | 0.4 (1.11) | 0.2 (0.46) | 0.3 (0.86)
  Ability To Eat (Day 5): number analyzed (Participants) | 39 | 41 | 27
  Ability To Eat (Day 5) | 0.3 (0.98) | 0.1 (0.36) | 0.3 (0.86)
  Ability To Deep Breath (Day 1): number analyzed (Participants) | 41 | 42 | 28
  Ability To Deep Breath (Day 1) | 1.5 (2.51) | 0.7 (1.27) | 1.5 (2.32)
  Ability To Deep Breath (Day 2): number analyzed (Participants) | 42 | 43 | 30
  Ability To Deep Breath (Day 2) | 1.2 (2.06) | 0.8 (1.43) | 1.1 (1.82)
  Ability To Deep Breath (Day 3): number analyzed (Participants) | 42 | 45 | 28
  Ability To Deep Breath (Day 3) | 1.4 (2.39) | 0.5 (1.06) | 0.7 (1.28)
  Ability To Deep Breath (Day 4): number analyzed (Participants) | 38 | 44 | 29
  Ability To Deep Breath (Day 4) | 1.1 (1.93) | 0.5 (0.90) | 0.7 (1.56)
  Ability To Deep Breath (Day 5): number analyzed (Participants) | 39 | 42 | 27
  Ability To Deep Breath (Day 5) | 0.8 (1.86) | 0.4 (0.86) | 0.4 (0.69)
  Ability To Cough (Day 1): number analyzed (Participants) | 40 | 44 | 28
  Ability To Cough (Day 1) | 4.4 (3.41) | 3.8 (3.10) | 5.7 (3.06)
  Ability To Cough (Day 2): number analyzed (Participants) | 41 | 43 | 30
  Ability To Cough (Day 2) | 4.4 (3.10) | 3.4 (2.61) | 5.0 (2.99)
  Ability To Cough (Day 3): number analyzed (Participants) | 42 | 45 | 27
  Ability To Cough (Day 3) | 3.9 (3.08) | 2.9 (2.28) | 4.5 (3.12)
  Ability To Cough (Day 4): number analyzed (Participants) | 38 | 44 | 29
  Ability To Cough (Day 4) | 3.2 (2.76) | 2.3 (2.02) | 3.5 (2.97)
  Ability To Cough (Day 5): number analyzed (Participants) | 38 | 42 | 27
  Ability To Cough (Day 5) | 3.0 (2.77) | 2.2 (1.97) | 3.1 (2.71)

ADVERSE EVENTS:
Time Frame: Through study completion, approximately 14 days
Groups:
- Group 1: SABER-Bupivacaine: 2.5 mL SABER-Bupivacaine /Once
  SABER-Bupivacaine: Injectable Extended Release Solution; 2.5 mL SABER-Bupivacaine(330 mg)/Once
- Group 2: SABER-Bupivacaine: 5.0 mL SABER-Bupivacaine /Once
  SABER-Bupivacaine: Injectable Extended Release Solution; 5.0 mL SABER-Bupivacaine (660 mg) /Once
Arm/Group | Group 1: SABER-Bupivacaine | Group 2: SABER-Bupivacaine | Group 3: SABER-Placebo
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/47 | 0/32
Serious Adverse Events (participants affected / at risk) | 3/44 | 2/47 | 1/32
Other Adverse Events (participants affected / at risk) | 44/44 | 44/47 | 31/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: SABER-Bupivacaine (N=44) | Group 2: SABER-Bupivacaine (N=47) | Group 3: SABER-Placebo (N=32)
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 1
Syncope vasovagal (Nervous system disorders) | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: SABER-Bupivacaine (N=44) | Group 2: SABER-Bupivacaine (N=47) | Group 3: SABER-Placebo (N=32)
Bradycardia (Cardiac disorders) | 9 | 12 | 7
Tinnitus (Ear and labyrinth disorders) | 3 | 6 | 5
Constipation (Gastrointestinal disorders) | 17 | 13 | 18
Nausea (Gastrointestinal disorders) | 14 | 9 | 10
Vomiting (Gastrointestinal disorders) | 3 | 1 | 2
Application site discoloration (General disorders) | 10 | 11 | 6
Pyrexia (General disorders) | 1 | 2 | 2
Incision site infection (Infections and infestations) | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0
Dizziness (Nervous system disorders) | 14 | 11 | 10
Dysgeusia (Nervous system disorders) | 6 | 5 | 5
Headache (Nervous system disorders) | 11 | 9 | 7
Paraesthesia (Nervous system disorders) | 9 | 5 | 2
Somnolence (Nervous system disorders) | 20 | 18 | 16
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 11 | 7
Hypotension (Vascular disorders) | 3 | 2 | 3
Incision site oedema (Injury, poisoning and procedural complications) | 3 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes